CLINICAL TRIAL: NCT04335838
Title: Age, Traumatic Brain Injury and Injury Severity as Independent Risk Factors for In-Hospital Mortality in Polytrauma Patients. Experiences From a Level I Trauma Center.
Brief Title: Age, Traumatic Brain Injury and Injury Severity as Independent Risk Factors for In-Hospital Mortality in Polytrauma Patients.
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Valerie Weihs, Principle Investigator, Medical University of Vienna
Other Study IDs: 1816/2016
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Polytrauma; Traumatic Brain Injury
Keywords: prognostic factors; New Berlin Definition; Polytrauma
MeSH Terms: conditions — Multiple Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polytrauma Patients: Patients with an ISS >16 points, an AIS >3 in one body region and at least 2 different body regions affected were included.
  Interventions: Other: retrospective analysis

INTERVENTIONS:
Other: retrospective analysis — The investigators retrospectively analyzed the outcome and possible prognostic factors in polytrauma patients.

SUMMARY:
In this study patients who were admitted to our hospital with critical injuries were enrolled retrospectively from January 2012 to December 2015. Patients with an ISS>16 points, an AIS >3 in one body region and at least 2 different body regions affected were included. Possible prognostic factors were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ISS >16 points
* AIS >3 in one body region
* at least 2 body regions affected

Exclusion Criteria:

* patients younger than 18 years of age
* isolated traumatic brain injury
* minor injuries (AIS <3 or ISS <16 points)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of polytrauma patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality in polytrauma patients. | January 1, 2012 to December 31, 2015

SECONDARY OUTCOMES:
Possible prognostic factors influencing the outcome of polytrauma patients. | Januar 1, 2012 to December 31, 2015
  Evaluation of concomitant traumatic brain injury, resuscitation, injury severity and trauma mechanisms in polytrauma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Traumatology, Vienna, Austria